CLINICAL TRIAL: NCT02416427
Title: A Phase II, Randomized, Non-comparative, Pre-surgical Study of Atorvastatin or Observation in Ki-67 Positive, TAZ-expressing Early Breast Cancer Patients (TRINACRIA Trial)
Brief Title: Targeting the Hippo Transducer TAZ in Breast Cancer With Statins
Acronym: TRINACRIA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Dr. Marcello Maugeri-Saccà, MD, PhD, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 637/15
Record Dates: First submitted 2015-04-02; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Breast Neoplasms
Keywords: Atorvastatin; TAZ; Hippo pathway; ki67
MeSH Terms: conditions — Breast Neoplasms | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Atorvastatin 80 mg/day for 3 weeks
  Interventions: Drug: Atorvastatin
- Arm B (No Intervention): Observation

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin will be administered at 80 mg/day for 3 weeks in the time window between diagnostic biopsy and curative surgery
  Arms: Arm A

SUMMARY:
This pre-surgical, window-of-opportunity study is designed to investigate whether atorvastatin reduces the proliferation marker Ki-67 via modulation of the Hippo transducer TAZ.

ELIGIBILITY:
Inclusion:

* Signed written informed consent
* Female aged >18 years and <75 years at the time of the enrolment
* Histologically confirmed Breast Cancer (BC) independently on the intrinsic subtype
* Stage I-IIa BC patients candidate for elective surgery
* BC expressing Ki-67 ≥ 15% and TAZ > 10% in diagnostic core biopsies
* Adequate baseline organ function
* Negative pregnancy test

Exclusion:

* Previous systemic therapy including chemotherapy, hormone therapy and targeted agents
* Administration of an investigational drug prior to enrolment
* History of another malignancy, except for a history of completely resected non-melanoma skin cancer or successfully treated cervical in situ carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status ≥2
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome and asymptomatic gallstones)
* Serious cardiac illness or medical conditions including but not confined to: history of documented congestive heart failure (CHF) or systolic dysfunction (LVEF <50%); high-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV-block, supraventricular arrhythmias which are not adequately controlled); angina pectoris requiring antianginal medication; clinically significant valvular heart disease; evidence of transmural infarction on ECG; poorly controlled hypertension (e.g. systolic >180mm Hg or diastolic >100mm Hg)
* Have a concurrent disease or condition that may interfere with study participation, or any serious medical disorder that would interfere with the subject's safety (for example, active or uncontrolled infection or any psychiatric condition prohibiting understanding or rendering of informed consent)
* Current or recent therapy with statins for hypercholesterolemia or other lipid-lowering drugs
* Current or recent therapy with glucose-lowering drugs for diabetes
* Current or recent therapy with strong CYP3A4 inhibitors (e.g., clarithromycin, HIV protease inhibitors, itraconazole) given potential interactions with atorvastatin
* Current or recent therapy with gemfibrozil or other fibrates given potential interactions with atorvastatin.
* Patients who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ki-67 reduction below the 15% (marker response). | 4 weeks

SECONDARY OUTCOMES:
• Decreased TAZ expression | 4 weeks
  Reduced TAZ expression evaluated by IHC when comparing pre- and post-treatment samples. Staining intensity will be graded on a four-grade scale (0: negative, 1: weak, 2: moderate, 3: strong). The final score will be obtained by considering staining intensity, percentage of expressing cells, and localization (nuclear versus cytoplasmic)
Pathway inhibition | 4 weeks
  Decreased expression of TAZ targets (AXL and CTGF) and Atorvastatin target (HMGCoAR) evaluated by IHC when comparing pre- and post-treatment samples. Staining intensity for all the molecular endpoints analyzed will be graded on a four-grade scale (0: negative, 1: weak, 2: moderate, 3: strong).